CLINICAL TRIAL: NCT05004155
Title: Twenty Four Hour Ambulatory pH & Impedance Testing: Normative Data for Indian Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Rakesh Kalapala, Doctor, Asian Institute of Gastroenterology, India
Other Study IDs: AIG/IEC-BH&R 11/03 2021-01
Record Dates: First submitted 2021-08-04; First posted 2021-08-13 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Esophageal Diseases; Esophagitis; Reflux Disease
Keywords: esophageal diseases; normative data; Reflux disease
MeSH Terms: conditions — Esophageal Diseases; Esophagitis; Gastroesophageal Reflux | interventions — Hydrogen-Ion Concentration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 24 hour pH & impedance monitoring — 24 hour pH impedance monitoring will be done on healthy subjects so that normative data specific to indian population can be generated.

SUMMARY:
GERD is common in Indian population and the normative data which is used to diagnose & manage GERD and its complications are based on western data which is not validated in the Indian population. Although normative data is available for commonly used twenty-four impedance-pH parameters, their global application has limitations, stemming from use of small healthy volunteer cohorts from few countries for normative data. At present, there is no normative data for twenty-four hours impedance-pH monitoring in Indian population. The aim of this study is to obtain a new set of normal values specific for the Indian population.

DETAILED DESCRIPTION:
1. INTRODUCTION Ambulatory impedance-pH monitoring is well established in the investigation of oesophageal symptoms suspicious of gastro-oesophageal reflux disease (GERD), and may be of particular value where symptoms persist or do not improve with empiric GERD treatment trials or GERD management, or where the diagnosis of GERD is inconclusive. Although normal values are available for commonly used impedance-pH parameters, their global application has limitations, stemming from use of small healthy volunteer cohorts from one or two countries for normative data. Further, significant technical limitations in analysis exist, such as inclusion of pH drops from meals/artefacts and inconsistent rules for identification of impedance reflux events, leading to large inter-reviewer variability. Several measurement systems are used for impedance-pH monitoring worldwide. Despite regional differences in prevalence of GERD phenotypes, symptomatic profiles and GERD complications, the same impedance-pH threshold values are used to define normality by these measurement systems. It remains unclear if measurements obtained using different systems or across world regions are comparable, especially since automated analysis provided by impedance-pH systems suffers from significant overcall of reflux episodes. Accurate identification and quantification of acid and non-acid reflux episodes on impedance-pH monitoring is important for precise calculation of oesophageal acid exposure time (AET), for reflux-symptom association analysis, and for evaluation of clearance mechanisms such as the postreflux swallow induced peristaltic wave (PSPW). Both reflux episodes and PSPW need to be reliably identified and recorded, for correct calculation of the PSPW index. Baseline impedance from impedance-pH monitoring can provide a measure of oesophageal mucosal integrity. Baseline impedance during the nocturnal supine period has been shown to be higher in healthy subjects and patients with functional heartburn and lower in patients with reflux disease. We aimed to obtain a new set of normal values for impedance- pH monitoring based on consensus analysis of impedance pH studies performed using different hardware/software systems from a large worldwide cohort of healthy asymptomatic subjects.
2. RATIONALE Although normal values are available for commonly used impedance-pH parameters, their global application has limitations, stemming from use of small healthy volunteer cohorts from one or two countries for normative data. At present, there is no normative data for impedance-pH monitoring in Indian population. The aim of this study is to obtain a new set of normal values specific for the Indian population.
3. STUDY OBJECTIVES 3a. Primary objective - To establish normative data for impedance-pH monitoring in Indian population.
4. STUDY POPULATION- 50 healthy asymptomatic subjects
5. DESIGN AND DURATION OF THE STUDY- It will be a observational prospective study. The study duration will be till completion of data collection for 50 subjects.

6a. SUBJECT RECRUITMENT - Healthy volunteers

6b. RANDOMIZATION AND BLINDING- Not applicable

6c. STUDY METHODS- This observational study will be conducted among 50 patients of both sexes after obtaining ethical clearance from institutional human ethical committee. Study participants will be of the age more than 18 years. Exclusion criteria will consist of thoracic or digestive foregut surgery, alcohol consumption >40 g/day, use of medications that alter intragastric acidity or oesophageal motility, as well as history of diabetes mellitus, neurological disorders or other chronic gastrointestinal disease.

6d. STUDY PROCEDURE- After at least 6 hours of fasting, a catheter will be placed through the nasal passage, and then swallowed into the esophagus with drinks of water. The other end of the catheter will be taped to cheek, wrapped over ear, and attached to a small data recorder that the subject will wear at waist level, held by a strap over the shoulder. Subject will be able to swallow, talk, and breathe without any difficulty during the test. Placement of the catheter will take about 10 minutes. One pH electrode will be positioned 5 cm proximal to the manometrically identified lower oesophageal sphincter (LES), and six impedance channels with their midpoint located 3, 5, 7, 9, 15 and 17 cm proximal to the LES. During the recording period, subjects will be encouraged to continue with their usual daily activities and meals. Subjects will be asked to keep a diary during the testing, including every time you eat, drink, or take medicines, and how long that lasts, when you lie down and get up, and each and every time you have a symptom of interest (like heartburn, regurgitation, cough, sore throat, etc.). Subject cannot take a shower or bath while wearing the monitor. Suject will return next day to have the catheter removed and to turn in the diary. Removing the catheter takes less than one minute. The total duration of catheter placement will be 24 hours. The equipment used will be pH monitoring catheter (Alacer, Brazil).

6e. METHODS OF ASSESSMENT- All tracings will be initially checked, and excluded if they had technical artefacts, marked oesophageal symptoms or antireflux medication intake. During the subsequent analysis process, tracings will be excluded if they fulfilled criteria for behavioural disorders (aerophagia, supragastric belching and rumination), low mean nocturnal baseline impedance (MNBI) in all impedance channels suspicious for eosinophilic oesophagitis (EoE) and hiatal hernia larger than 2 cm (in those with available HRM). All tracings will be analysed by four individuals, each with experience in reviewing >300 impedance-pH studies annually. Reviewers will initially apply automated analysis, followed by manual review of each identified reflux episode and PSPW for accuracy, as well as manual addition of missed events identified within the time window of 3 min used to edit the reflux events detected by automated analysis, with two reviewer consensus for each retained episode. The analysis process will consist of: (1) editing of pH drops (to exclude artefacts and meal/drink induced pH drops). Slow pH drifts without impedance reflux were included for calculation of total AET but were not considered separate reflux episodes. (2) Identification of impedance reflux events and PSPW using strict pre-established criteria and (3) measurement of distal MNBI. After manual editing, the following parameters will be considered for normative data: total, upright and supine AET, number of reflux events (total, acid and non-acid), PSPW index and MNBI at 3 and 5 cm above the LES.

6f. STOPPING OR DISCONTINUATION CRITERIA- Not applicable

7. OUTCOME MEASURES 7a. Primary - To establish normative data for impedance-pH monitoring in Indian population.

There are no secondary objectives.

8. STATISTICAL ANALYSIS- Data will be expressed as median and percentile values (5th, 25th, 75th and 95th percentiles). Depending on normality of distribution, we will use either paired Student's t-test or Mann-Whitney U test for paired comparison. Likewise, we will use one way analysis of variance with Tukey test or Kruskal-Wallis, followed by Dunn's test as appropriate. Upper limit of normal will be defined as the 95th percentile of normal values. For PSPW index and MNBI thresholds, we will use the 5th and 25th percentile values. P≤0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individual > 18 years of age
* Not on any acid lowering drug from at least 7 days.

Exclusion Criteria:

* Thoracic or digestive foregut surgery,
* Alcohol consumption >40 g/day,
* Use of medications that alter intragastric acidity or oesophageal motility
* History of diabetes mellitus,
* Neurological disorders
* Chronic gastrointestinal disease
* Any subject with upper GI symptoms like pain, burning, belching, bloating, dysphagia & aerophagia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will enroll only healthy asymtomatic subjects, so that normative data can be generated.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Normative values for impedance-pH monitoring in healthy Indian population. | six months
  There is no normative data for impedance-pH monitoring specific to indian population. The study aims to generate a reference value for the same by enrolling healthy individuals.

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh kalapala, MBBS, MD, DM, Study Director — Senior Consultant; Pradev Inavolu, Principal Investigator — Consultant; Hardik Rughwani, Principal Investigator — Consultant
Locations (1):
- AIG Hospitals, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD.

REFERENCES:
- [Result] Sifrim D, Roman S, Savarino E, Bor S, Bredenoord AJ, Castell D, Cicala M, de Bortoli N, Frazzoni M, Gonlachanvit S, Iwakiri K, Kawamura O, Krarup A, Lee YY, Soon Ngiu C, Ndebia E, Patcharatraku T, Pauwels A, Perez de la Serna J, Ramos R, Remes-Troche JM, Ribolsi M, Sammon A, Simren M, Tack J, Tutuian R, Valdovinos M, Xiao Y, Zerbib F, Gyawali CP. Normal values and regional differences in oesophageal impedance-pH metrics: a consensus analysis of impedance-pH studies from around the world. Gut. 2020 Oct 9:gutjnl-2020-322627. doi: 10.1136/gutjnl-2020-322627. Online ahead of print. PMID 33037054
- [Result] Roman S, Gyawali CP, Savarino E, Yadlapati R, Zerbib F, Wu J, Vela M, Tutuian R, Tatum R, Sifrim D, Keller J, Fox M, Pandolfino JE, Bredenoord AJ; GERD consensus group. Ambulatory reflux monitoring for diagnosis of gastro-esophageal reflux disease: Update of the Porto consensus and recommendations from an international consensus group. Neurogastroenterol Motil. 2017 Oct;29(10):1-15. doi: 10.1111/nmo.13067. Epub 2017 Mar 31. PMID 28370768
- [Result] Zerbib F, des Varannes SB, Roman S, Pouderoux P, Artigue F, Chaput U, Mion F, Caillol F, Verin E, Bommelaer G, Ducrotte P, Galmiche JP, Sifrim D. Normal values and day-to-day variability of 24-h ambulatory oesophageal impedance-pH monitoring in a Belgian-French cohort of healthy subjects. Aliment Pharmacol Ther. 2005 Nov 15;22(10):1011-21. doi: 10.1111/j.1365-2036.2005.02677.x. PMID 16268977
- [Result] Shay S, Tutuian R, Sifrim D, Vela M, Wise J, Balaji N, Zhang X, Adhami T, Murray J, Peters J, Castell D. Twenty-four hour ambulatory simultaneous impedance and pH monitoring: a multicenter report of normal values from 60 healthy volunteers. Am J Gastroenterol. 2004 Jun;99(6):1037-43. doi: 10.1111/j.1572-0241.2004.04172.x. PMID 15180722